CLINICAL TRIAL: NCT00681265
Title: A Randomized, Masked Exploratory Trial Comparing the Effect of Two Different Over-the-Counter Artificial Tear Preparations on Tear Film Break-up Time
Brief Title: Tear Film Break-up Time After Instillation of Artificial Tears
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Calm Water Therapeutics LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: ET-001
Record Dates: First submitted 2008-05-19; First posted 2008-05-21 (Estimated); Results first posted 2012-10-26 (Estimated); Last update posted 2012-10-26 (Estimated); Status verified 2012-10

CONDITIONS: Keratoconjunctivitis Sicca
Keywords: ocular lubricants
MeSH Terms: conditions — Keratoconjunctivitis Sicca | interventions — Glycerol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- glycerin (Experimental): One eye will randomly receive a single instillation of one drop of a new formulation of an artificial tear containing glycerin 1% as an active with polylysine-graft-polyethylene glycol as an excipient.
  Interventions: Drug: glycerin
- polyethylene glycol 400/propylene glycol (Active Comparator): The other eye will receive a single instillation of one drop of an artificial tear with propylene glycol (0.3%) and polyethylene glycol (0.4%) as active ingredients with hydroxypropyl-guar as a gelling agent.
  Interventions: Drug: polyethylene glycol 400/propylene glycol

INTERVENTIONS:
Drug: glycerin — Eye drop with active agent glycerin 1%, new topical ophthalmic formulation with polylysine-graft-polyethylene glycol as an excipient, single instillation.
  Other Names: Eyeon Protect(TM)
  Arms: glycerin
Drug: polyethylene glycol 400/propylene glycol — Eye drop with the active agents polyethylene glycol 400 0.4% /propylene glycol 0.3%, topical ophthalmic formulation, single instillation
  Other Names: Systane(R)
  Arms: polyethylene glycol 400/propylene glycol

SUMMARY:
This study is an exploratory trial evaluating the tear film break-up time after a single eye drop instillation of over-the-counter artificial tears. The primary hypothesis is that tear film break up time will be greater for test than control eye.

DETAILED DESCRIPTION:
Subjects with varying degrees of dry eye syndrome were enrolled in a randomized, controlled, double masked, single site study. A new formulation of an artificial tear containing glycerin 1% as an active with polylysine-graft-polyethylene glycol as an excipient was compared against a leading commercial product with propylene glycol (0.3%) and polyethylene glycol (0.4%) as active ingredients with hydroxypropyl-guar as a gelling agent. The primary outcome was a comparison of tear film stability after eye drop instillation.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* symptoms of dry eye
* no other history of ophthalmic problems

Exclusion Criteria:

* Use of any ocular lubricant or ointment in the past 36 hours
* use of contact lenses or excessive eye lid cosmetics on the study day

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2008-06; Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James V. Aquavella, MD, Principal Investigator — University of Rochester Eye Institute
Locations (1):
- University of Rochester Eye Institute, Rochester, New York, United States

REFERENCES:
- [Background] Nichols JJ, Nichols KK, Puent B, Saracino M, Mitchell GL. Evaluation of tear film interference patterns and measures of tear break-up time. Optom Vis Sci. 2002 Jun;79(6):363-9. doi: 10.1097/00006324-200206000-00009. PMID 12086302
- [Background] Ousler GW, Michaelson C, Christensen MT. An evaluation of tear film breakup time extension and ocular protection index scores among three marketed lubricant eye drops. Cornea. 2007 Sep;26(8):949-52. doi: 10.1097/ICO.0b013e3180de1c38. PMID 17721294
- [Background] Cho P, Douthwaite W. The relation between invasive and noninvasive tear break-up time. Optom Vis Sci. 1995 Jan;72(1):17-22. doi: 10.1097/00006324-199501000-00004. PMID 7731650

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Dates: 5/18/2008 to 8/30/2008. Single site: Flaum Eye Institute at the University of Rochester.
Groups:
- Glycerin Eye Drop / PEG 400 and Propylene Glycol Eye Drop: One eye will randomly receive a single instillation of one drop of a new formulation of an artificial tear containing glycerin 1% as an active with polylysine-graft-polyethylene glycol as an excipient. The other eye will receive a single instillation of one drop of an artificial tear with propylene glycol (0.3%) and polyethylene glycol (0.4%) as active ingredients with hydroxypropyl-guar as a gelling agent.
Period: Overall Study
Arm/Group | Glycerin Eye Drop / PEG 400 and Propylene Glycol Eye Drop
Started | 16
Completed | 16
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Glycerin Eye Drop / PEG 400 and Propylene Glycol Eye Drop
Number analyzed (Participants) | 16
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 16
  >=65 years | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 44.5 (10.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 6
Region of Enrollment [Number; unit: participants]
  United States | 16

OUTCOME MEASURES:

1. Primary Outcome: Noninvasive Tear Film Break-up Time
Description: State-of-the-art methodology to assess tear stability.
Time Frame: 15 minutes after eye drop instillation
Population: Study N determined empirically by PI.
Measure: Mean (Standard Deviation); unit: seconds
Groups:
- New Formulation of Glycerin 1% Eye Drop: One eye will randomly receive a single instillation of one drop of a new formulation of an artificial tear containing glycerin 1% as an active with polylysine-graft-polyethylene glycol as an excipient.
- Propylene Glycol and PEG 400 Eye Drop: The other eye will receive a single instillation of one drop of an artificial tear with propylene glycol (0.3%) and polyethylene glycol (0.4%) as active ingredients with hydroxypropyl-guar as a gelling agent.
Arm/Group | New Formulation of Glycerin 1% Eye Drop | Propylene Glycol and PEG 400 Eye Drop
Number analyzed (Participants) | 16 | 16
seconds | 14.67 (27.21) | 7.4 (30.30)

2. Secondary Outcome: Fluorescein Tear Film Break-up Time
Description: Standard clinical assessment methodology for assessing tear stability.
Time Frame: 120 minutes after eye drops instillation
Population: Study N determined empirically by PI.
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | New Formulation of Glycerin 1% Eye Drop | Propylene Glycol and PEG 400 Eye Drop
Number analyzed (Participants) | 16 | 16
seconds | 11.13 (12.08) | 6.21 (4.86)

ADVERSE EVENTS:
Arm/Group | New Formulation of Glycerin 1% Eye Drop | Propylene Glycol and PEG 400 Eye Drop
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/16
Other Adverse Events (participants affected / at risk) | 0/16 | 0/16

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No